CLINICAL TRIAL: NCT00491192
Title: Normothermia in Patients With Acute Cerebral Damage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1575
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-06

CONDITIONS: Traumatic Brain Injury; Subarachnoid Hemorrhage
Keywords: Fever; Acute cerebral damage; Normothermia; Diclofenac; ICU; Outcome; Intracranial pressure; Cerebral perfusion pressure; Traumatic brain injury; Subarachnoid hemorrhage
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Fever | interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Diclofenac

SUMMARY:
The purpose of our study is to verify wherever normothermia (achieved with diclofenac administration) may improve intracranial pressure control and may limit secondary cerebral damage thus positively influencing outcome in patients with acute cerebral damage admitted to ICU.

DETAILED DESCRIPTION:
Pyrexia can exacerbate ischemic neuronal damage and physiological dysfunction after traumatic brain injury and subarachnoid hemorrhage.Fever also represent an important issue occurring in 78% of patients with acute cerebral damage admitted to intensive care unit (ICU). For those patients, normothermia is actually recommended in order to reduce secondary cerebral damage and to control intracranial pressure, that are known to worsen long term prognosis. Our primary endpoint is to maintain normothermia in patients with acute cerebral damage (axillary temperature < 38°C or internal temperature < 38,8°C) administering diclofenac. We will also investigate the corresponding behaviour of intracranial pressure and cerebral perfusion pressure.

Comparison(s): We will compare two different doses of subcutaneous diclofenac (0,35 mg/kg - 1/3 a vial - vs 0,5 mg/Kg - 1/2 vial) to continuous intravenous of 0,48 mg/kg diclofenac for 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe traumatic injury or subarachnoid hemorrhage in coma (GCS<8), intubated, mechanically ventilated with intracranial pressure (ICP) and invasive arterial pressure monitoring

Exclusion Criteria:

* Know adverse reactions with NSAI
* Platelets count < 20,000/dl
* Gastric or duodenal ulceration in active phase
* Hepatic insufficiency, cirrhosis or previous liver transplant
* Acute or chronic renal insufficiency
* Coronary insufficiency, acute myocardial infarct in the previous 6 month
* Barbiturate coma
* Patients in therapy with acetylsalicylic acid, lithium, digoxin, methotrexate and cyclosporin.
* Known or suspected pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-06; Study Completion 2009-06

PRIMARY OUTCOMES:
Maintenance of normothermia | within 14 days from ICU admission

SECONDARY OUTCOMES:
Behaviour of intracranial pressure and cerebral perfusion pressure. Influence on six month outcome. | Within 14 days from ICU admission/Six months

CONTACTS AND LOCATIONS:
Overall Officials: Nino Stocchetti, MD, Study Director — Ospedale Maggiore Policlinico Mangiagalli e Regina Elena
Locations (1):
- Fondazione Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, Milan, Italy